CLINICAL TRIAL: NCT06170346
Title: The Effect of Topical Agents With Various Antioxidant Containts on Photodamage Skin Induced by Ultraviolet B Radiation
Brief Title: Effect of Topical Agents With Various Antioxidant Containts on Photodamage Skin Induced
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DV-202309.01
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Photodamaged Skin
Keywords: Antioxidants
MeSH Terms: interventions — Antioxidants

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Antioxidant (Experimental): 30 drops of topical antioxidants (Gluconolactone 4%, Hyaluronic acid 0,01%, Allantoin 0,1%, Ferulic acid 3%, Acetyl heptapeptide 0,001%, Silver vine extract 1%, Ectoine 0,01%, Hydroxyectoine 0,01%, and vehicle) will be applied on tested area on each participant for four consecutive days. On the fifth day, the subject will be irradiated on the tested area. After irradiation, erythema intensity and skin biopsy will be taken. Furthermore, skin tissue will be stained to see sunburn cells and assesses the expression of MMP-9, Thymine Dimer, and p-53 by immunohistochemistry.
  Interventions: Combination Product: Antioxidants
- Vehicle (Placebo Comparator): 30 drops of topical vehicle (Aqua, Dipropylene glycol, Hydroxypropyl cyclodextrin, Polydextrose, 1,2-hexanediol, Butylene glycol, Propanediol, Caprylhydroxamic acid, Ethylhexylglycerin, Xanthan gum, Benzyl alcohol, Glyceryl caprylate, and Benzoic acid) will be applied on tested area on each participant for four consecutive days. On the fifth day, the subject will be irradiated on the tested area. After irradiation, erythema intensity and skin biopsy will be taken. Furthermore, skin tissue will be stained to see sunburn cells and assesses the expression of MMP-9, Thymine Dimer, and p-53 by immunohistochemistry.
  Interventions: Combination Product: Vehicle
- Control (No Intervention): Skin without intervention and irradiation. Skin biopsy will be taken as a control. Skin tissue will be stained to see sunburn cells and assesses the expression of MMP-9, Thymine Dimer, and p-53 by immunohistochemistry.

INTERVENTIONS:
Combination Product: Antioxidants — 30 drops of topical antioxidants (Gluconolactone 4%, Hyaluronic acid 0,01%, Allantoin 0,1%, Ferulic acid 3%, Acetyl heptapeptide 0,001%, Silver vine extract 1%, Ectoine 0,01%, Hydroxyectoine 0,01%, and vehicle) will be applied on tested area on each participant for four consecutive days.
  Arms: Antioxidant
Combination Product: Vehicle — 30 drops of topical vehicle (Aqua, Dipropylene glycol, Hydroxypropyl cyclodextrin, Polydextrose, 1,2-hexanediol, Butylene glycol, Propanediol, Caprylhydroxamic acid, Ethylhexylglycerin, Xanthan gum, Benzyl alcohol, Glyceryl caprylate, and Benzoic acid) will be applied on tested area on each participant for four consecutive days.
  Arms: Vehicle

SUMMARY:
Ultraviolet (UV) irradiation of the skin leads to acute inflammatory reactions such as erythema, sunburn, and chronic reactions, including premature skin aging and skin tumors. UV irradiation is a potent generator of oxidative stress in the skin. Exposure of mammalian skin to UV increases the cellular levels of reactive oxygen species, which damages lipids, proteins, and nucleic acids in both epidermal and dermal cells and contributes to the sunburn reaction as well as photocarcinogenesis and photoaging. In this study, the effects of a topical antioxidant on attenuating the harmful effects of UV irradiation on normal healthy volunteers were studied using biomarkers of skin damage. This study confirms the protective role of a unique mixture of antioxidants on human skin from the harmful effects of UV irradiation. We propose that antioxidant mixture will complement and synergize with sunscreens in providing photoprotection for human skin.

DETAILED DESCRIPTION:
Photoprotection is an effort made to reduce the detrimental effects of Reactive Oxygen Species (ROS) on the skin due to UVB exposure. Photoprotection consists of primary and secondary. Lifestyle modification, physical photoprotection and sunscreen use are parts of primary photoprotection. Secondary photoprotection is the use of agents or ingredients that serve to reduce the adverse effects of sunlight reaching the skin. Examples of secondary photoprotection are antioxidants. Antioxidants are compounds that in low levels react with oxidized substrates by providing electrons. These compounds can prevent and neutralize the negative impact of ROS on the skin due to UVB exposure, one of which is minimizing photoaging. UVB exposure can produce ROS that trigger erythema in subjects, the formation of DNA damage in the form of thymine dimers, the discovery of sunburn cells and can activate p53, and MMP-9 enzymes. Acute photodamage is characterized by the formation of sunburn cells and chronically can lead to malignancy. Photoprotection can be used to reduce these effects. One of the photoprotection efforts is the use of antioxidants, which are secondary photoprotective agents that prevent or repair skin damage caused by ROS. In previous studies, topical ingredients containing vitamin C, vitamin E, and ferulic acid have a photoprotective effect against UVB-induced skin photodamage characterized by decreased expression of thymine dimer and p53 in the skin. Various studies on the combined effects of antioxidant ingredients are still being developed. Currently, there is no research on the effect of topical ingredients containing various antioxidants, namely gluconolactone, hyaluronic acid, allantoin, ferulic acid, acetyl heptapeptide, silver vine extract, ectoine, and hydroxyectoine on skin photodamage. For this reason, it is necessary to conduct research on the effects of topical ingredients containing various antioxidants on the expression of thymine dimer and p53 in UVB-induced skin compared to vehiculum.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-60 years.
* Skin types III and IV according to Fitzpatrick.
* Normal back skin.

Exclusion Criteria:

* Pregnant and lactating women.
* History of photodermatosis, skin malignancies, skin diseases that can be exacerbated by light.
* History of sun exposure to the back area in the past two weeks.
* History of applying and taking antioxidants containing gluconolactone, hyaluronic acid, allantoin, ferulic acid, acetyl heptapeptide, silver vine extract, ectoine, and hydroxyectoine in the past 12 weeks.
* History of taking photosensitizer drugs (malaria drugs, analgesics, antidepressants, systemic fungal drugs, chemotherapy) in the past eight weeks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Erythema intensity | 1 day
  Assessment of the erythema intensity using a spectrophotometer
Sunburn cells | 1 day
  Assessment of sunburn cells numbers in epidermis from skin tissue stained using Hematoxylin Eosin.
MMP-9 expression | 1 day
  Assessment of MMP-9 expression in epidermis from skin tissue stained using Immunohistochemistry.
p53 expression | 1 day
  Assessment of p53 expression in epidermis from skin tissue stained using Immunohistochemistry.
Thymine dimer expression | 1 day
  Assessment of thymine dimer expression in epidermis from skin tissue stained using Immunohistochemistry.

CONTACTS AND LOCATIONS:
Overall Officials: Reti Hindritiani, M.D., Ph.D, Principal Investigator — Padjadjaran University
Locations (1):
- Hasan Sadikin General Hospital, Bandung, West Java, Indonesia